CLINICAL TRIAL: NCT00960336
Title: Multicenter Study of PEGylated Liposomal Doxorubicin in Geriatric Oncology - Metastatic Breast Cancer - First-line Treatment PEGylated Liposomal Doxorubicin in Patients Older Than 70 Years, Breast Cancer Metastasis
Brief Title: Doxorubicin Hydrochloride Liposome as First-Line Therapy in Treating Older Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000633600; ARCAGY-DOGMES; ARCAGY-GINECO-BR106; INCA-RECF0511; EUDRACT-2007-002736-28; SCHER-ARCAGY-DOGMES
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Breast Cancer
Keywords: HER2-negative breast cancer; recurrent breast cancer; stage IV breast cancer; invasive ductal breast carcinoma; invasive lobular breast carcinoma
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal, Breast; Carcinoma, Lobular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm (Experimental)
  Interventions: Drug: pegylated liposomal doxorubicin hydrochloride

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin hydrochloride liposome, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well doxorubicin hydrochloride liposome works as first-line therapy in treating older women with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the effectiveness of pegylated liposomal doxorubicin hydrochloride, in terms of objective response rate, in elderly women with metastatic breast cancer.

Secondary

* Determine the feasibility of this drug in these patients.
* Evaluate chemotherapy-induced toxicities in these patients.
* Assess the disease-free survival and overall survival of these patients.
* Study the geriatric covariates.
* Assess the covariates predictive of the hematopoietic reserve and the risk of febrile neutropenia in these patients.

OUTLINE: This is a multicenter study.

Patients receive pegylated liposomal doxorubicin hydrochloride IV over 60-90 minutes on day 1. Treatment repeats every 28 days for 6 courses in the absence of unacceptable toxicity or progressive disease.

After completion of study therapy, patients are followed up periodically for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive ductal or lobular adenocarcinoma of the breast

  * Metastatic disease as confirmed by ≥ 1 of the following:

    * Histology or cytology
    * Radiology
    * Elevated CA 15-3 levels
* No HER2/neu overexpression by IHC or FISH
* Measurable (≥ 10 mm) or evaluable disease

  * Bone lesions or isolated pleural effusion allowed
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Postmenopausal
* Life expectancy > 3 months
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* AST and ALT ≤ 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)
* Alkaline phosphatase ≤ 5 times ULN
* Bilirubin ≤ 2 times ULN
* Creatinine clearance ≥ 30 mL/min
* LVEF ≥ 50%
* No congestive heart failure or other uncontrolled cardiac disease
* No other malignancy within the past 5 years except for curatively treated carcinoma in situ of the cervix, urothelial in situ carcinoma, or basal cell cancer
* No prior hypersensitivity to anthracyclines
* No psychological, familial, social, or geographical reason that would preclude study follow-up
* No serious illness or physical or mental condition resulting in a permanent disability that may preclude successful treatment

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for metastatic disease
* Prior adjuvant chemotherapy allowed

  * No development of metastatic disease within 6 months after completion of adjuvant anthracycline-based chemotherapy
* No more than 300 mg/m² of prior doxorubicin hydrochloride or 600 mg/m² of prior epirubicin hydrochloride in the adjuvant setting
* More than 30 days since prior participation in another clinical trial

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 59 (Actual)
Dates: Start 2008-03; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Response rate | 3 and 6 cures

CONTACTS AND LOCATIONS:
Overall Officials: Laure Chauvenet, MD, Principal Investigator — Hotel Dieu de Paris
Locations (1):
- Hotel Dieu de Paris, Paris, France

REFERENCES:
- [Derived] Falandry C, Brain E, Bonnefoy M, Mefti F, Jovenin N, Rigal O, Guillem O, El Kouri C, Uwer L, Abadie-Lacourtoisie S, Cretin J, Jacquin JP, Paraiso D, Freyer G. Impact of geriatric risk factors on pegylated liposomal doxorubicin tolerance and efficacy in elderly metastatic breast cancer patients: final results of the DOGMES multicentre GINECO trial. Eur J Cancer. 2013 Sep;49(13):2806-14. doi: 10.1016/j.ejca.2013.04.027. Epub 2013 Jun 1. PMID 23735702